CLINICAL TRIAL: NCT05895929
Title: The Role of IL5 in Epithelial Cell Integrity
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00363909
Record Dates: First submitted 2023-05-12; First posted 2023-06-09 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyps; Chronic Rhinosinusitis (Diagnosis)
MeSH Terms: conditions — Disease | interventions — mepolizumab

STUDY DESIGN:
Intervention Model Description: Nasal epithelial cells will be exposed to defined doses of mepolizumab in vitro culture (Arm 1) or control media without mepolizumab (Arm 2)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mepolizumab treatment arm (Experimental): Nasal epithelial cells will be exposed in vitro to mepolizumab in culture.
  Interventions: Drug: Mepolizumab
- Control arm (No Intervention): Nasal epithelial cells will be exposed in vitro to media without mepolizumab in culture

INTERVENTIONS:
Drug: Mepolizumab — In vitro exposure of human nasal epithelial cells to mepolizumab
  Other Names: Nucala
  Arms: Mepolizumab treatment arm

SUMMARY:
The goal of this laboratory study is the examine the effect of mepolizumab drug on the health and function of the cells lining the human nasal airways in vitro cell culture derived from patients with chronic rhinosinusitis with nasal polyposis. The main questions the study aims to study are:

1. To see what mepolizumab does to suppress inflammation of the human cells.
2. To see what mepolizumab does to maintain barrier integrity of epithelial cells

DETAILED DESCRIPTION:
The investigators hypothesize that anti-IL5 treatment will promote epithelial cell function by inhibition of Type 1 and innate immune mediated inflammation and epithelial-mesenchymal transition resulting from IL5 induction.

Aim 1. To test the hypothesis that anti-IL5 therapy results in inhibition of epithelial cell dysfunction including epithelial derived inflammatory responses and barrier dysfunction, the investigators will examine the effect of in vitro anti-IL5 mepolizumab exposure of human primary nasal epithelial cells from chronic rhinosinusitis with nasal polyposis on Type 1, Type 2 and innate immune inflammatory markers, and markers of epithelial cell barrier function.

Aim 2. To examine the effect of mepolizumab to broadly modulate the expression of Type 2, Type 1, Type 3, and innate immune inflammatory gene responses in human nasal airway epithelial cells, the investigators will perform high throughput RNA sequencing on IL5 primed differentiated human primary nasal epithelial cells exposed to the presence and absence of mepolizumab in vitro cell culture which are derived from patients with chronic rhinosinusitis with nasal polyposis. These studies will provide an unbiased approach to identification of biomarkers resulting from anti-IL5 treatment.

ELIGIBILITY:
Inclusion Criteria:

* (1) sinonasal inflammation for greater than 12 weeks which include at least 2 of the following symptoms: nasal obstruction/congestion, nasal discharge (anterior or posterior), facial pressure/pain, reduction of sense of smell.
* (2) confirmation of the clinical symptoms by: (2a) CT scan evidence of paranasal sinus mucosal inflammation, and/or (2b) endoscopic exam evidence of purulence from the sinuses or ostiomeatal complex; and
* (3) presence of nasal polyps seen on endoscopic exam or sinus CT scan.

Exclusion Criteria:

* 1. Children under the age of 18 will be excluded due to:

  1. possible confounding diagnosis of cystic fibrosis and other non-Type 2 inflammatory etiologies that commonly presents with nasal polyps in the pediatric population.
  2. lack of complete pneumatization of the majority of paranasal sinuses
* 2. pregnant or lactating females,
* 3. prisoners,
* 4. mentally disabled
* 5. persons unable to give informed consent will be contemplated for inclusion.
* 6. disease secondary to a clearly defined anatomic process, such as facial trauma, and obstruction due to sinonasal neoplasm.
* 7. exposure to oral or systemic IV glucocorticoids within 2 weeks of surgery
* 8. exposure to immunomodulatory biologics will be excluded. These include, but are not limited to systemic treatment with biologics omalizumab, dupilumab, mepolizumab, benralizumab, reslizumab, or rituximab.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2023-09-05 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in Type 1 inflammatory markers (ng/mL) | 0 to 48 hours
  IL8 cytokine mRNA and protein expression
Change in Type 2 inflammatory markers (ng/mL) | 0 to 48 hours
  IL5 and thymic stromal lymphopoietin cytokine mRNA and protein expression
Change in Innate immune inflammatory markers (ng/mL) | 0 to 48 hours
  IL1 receptor mRNA and protein expression
Change in epithelial barrier function protein expression (ng/mL) | 0 to 48 hours
  E-cadherin
Change in epithelial integrity markers (staining intensity units) | 0 to 48 hours
  alpha-smooth muscle actin protein expression

CONTACTS AND LOCATIONS:
Overall Officials: Jean Kim, MD PhD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland